CLINICAL TRIAL: NCT03300128
Title: Evaluation of Incredible Years Parenting Program for Caregivers of Children with Autism
Brief Title: Incredible Years Program for Parents of Children with Autism
Acronym: IY-ASD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Sarah Dababnah, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00074617
Record Dates: First submitted 2017-09-22; First posted 2017-10-03 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2019-12

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; parenting; Incredible Years
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into a treatment group (IY-ASD parent training program) or comparison group ("Circle of Parents" parent support program). The 14-week parent groups will be offered twice per year. Once participants are enrolled in the study, they will complete a set of baseline measures (described in Section 5). The study coordinator will provide Dr. Dababnah a complete list of participants (unique identifiers only which do not contain identifiable information). Dr. Dababnah will randomize participants using a computer-generated randomization plan into either IY-ASD or "Circle of Parents" support group. While participants and the research team will not be blinded to group assignment, only the PI and her Research Assistant(s) at UMB will have access to the randomization plan. Dr. Dababnah and her team will review baseline measures for each period after individuals have been randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Incredible Years - ASD (Experimental): The intervention, The Incredible Years Parent Program for Autism Spectrum and Language Delays (IY-ASD; more information is here: http://www.incredibleyears.com/programs/parent/autism-spectrum-language-delays/) is a 14-week course that meets for 2 hours every week. Ideally, an IY-ASD group will be composed of approximately 10 parents and other primary caregivers of children who have autism.
  Interventions: Behavioral: Incredible Years - ASD
- Circle of Parents (Active Comparator): "Circle of Parents," the comparison condition, is an open parent support group led by a parent leader. (For more information, see http://circleofparents.org/). Participants are encouraged to share resources and other support both during groups, and between meetings.
  Interventions: Other: Circle of Parents

INTERVENTIONS:
Behavioral: Incredible Years - ASD — The IY-ASD intervention is designed for parents of children with autism spectrum disorder. The programs uses a mix of videos, collaborative brainstorming sessions, and role plays to deliver content on child-directed play and positive discipline practices.
  Other Names: Incredible Years
  Arms: Incredible Years - ASD
Other: Circle of Parents — "Circle of Parents" is an open parent support group led by a parent leader. Participants are encouraged to share resources and other support both during groups, and between meetings.
  Arms: Circle of Parents

SUMMARY:
Early intervention for children with Autism Spectrum Disorder (ASD), particularly with parent involvement, is beneficial for both children and their families. However, few interventions have been rigorously tested which explicitly address parent and family outcomes. This study will test the effectiveness of "The Incredible Years Parent Program for Autism Spectrum and Language Delays" (IY-ASD) program for parents of children with ASD ages 2-8 in a community-based setting, compared to a parent support program, "Circle of Parents." The investigators will assess parent stress, caregiver coping, child behavior, parenting practices of participants. In addition, the investigators will report on participants' satisfaction with IY-ASD, through parent interviews and satisfaction surveys.

DETAILED DESCRIPTION:
"The Incredible Years" refers to a suite of developmentally appropriate, group-based interventions targeting parenting, children, and teachers. IY-ASD is an adapted version of the Basic parent training program, which uses a simple and low-cost format to develop skills in problem-solving coping, stress management, and communication. "The Incredible Years" has decades of evidence pointing to improved levels of parent stress, depression, and coping skills, as well as decreased negative child outcomes such as aggressive behavior in a broad array of diverse populations. The program has been used extensively in the United Kingdom and Sweden. Cost-effectiveness analyses have been performed with positive results in England. "The Incredible Years" is based on attachment theory and social learning theory.The goals of "The Incredible Years" parent intervention - communication, problem-solving, and stress management - are critically important to this population. Parents with children with special needs tend to interact with teachers, healthcare professionals, and other adults more often than parents whose children do not have disabilities. Thus, building a strong foundation early to begin to problem solve, communicate effectively, and navigate healthcare and special education systems can reduce some stress the parent might experience in the future.

The Incredible Years Parent Program for Autism Spectrum and Language Delays (IY-ASD). IY-ASD will be delivered over a 14-week period. The current research aims to rigorously test IY-ASD in a community-based setting using a randomized design. The investigators will compare IY-ASD to a usual practice, a parent support group currently offered at Onslow County Partnership for Children, "Circle of Parents." "Circle of Parents" is an open group which is led by a parent leader. These groups generally meet weekly or biweekly. Participants are encouraged to share resources and other support both during groups, and between meetings. Free childcare and meals are also offered during "Circle of Parents" meetings. Using a randomized design, the investigators will evaluate a parent intervention for caregivers of children with Autism Spectrum Disorder (ASD), compared to a parent support group. Over a four-year period, the investigators seek to:

1. Recruit approximately 105 parents and other primary caregivers to participate in either an IY-ASD or "Circle of Parents" group;
2. Measure parenting stress, parent coping mechanisms, parenting practices, and child behavior of participants and their children, at baseline and posttest (pre- and post-intervention);
3. Compare outcomes of parents completing IY-ASD versus those in "Circle of Parents" group;
4. Evaluate changes in parent and child outcomes from post-intervention to 3-month follow-up in IY-ASD participants; and,
5. Elicit information from IY-ASD participants to assess satisfaction and improve future use of IY-ASD in the ASD population.

ELIGIBILITY:
Inclusion Criteria:

* Parent or primary caregiver of a child ages 2 to 8 with an autism spectrum disorder
* Must live in Onslow County or surrounding county

Exclusion Criteria:

* Parent is younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Change in child behavior | Change from baseline at 14 weeks and at 3 months
  Eyberg Child Behavior Inventory (ECBI) - This measure includes 36 items that assess typical problems reported by parents of conduct-disordered children. Items are rated on intensity and problem scales; the two subscales are combined for a composite score.
Change in parent stress | Change from baseline at 14 weeks and at 3 months
  Parenting Stress Index-Short Form (PSI-SF) - The PSI Short Form (PSI/SF) is a direct derivative of the Parenting Stress Index (PSI) full-length test. All 36 items on the Short Form are contained on the Long Form with identical wording and are written at a 5th-grade reading level, for parents of children 12 years and younger. The PSI/SF yields a Total Stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child.

SECONDARY OUTCOMES:
Change in coping mechanisms | Change from baseline at 14 weeks and at 3 months
  Brief COPE - This measures assesses several types of coping mechanisms used to address stress.
Change in parenting practices | Change from baseline at 14 weeks and at 3 months
  Parent Practices Inventory (PPI) - This questionnaire was adapted from the Oregon Social Learning Center's (OSLC) discipline questionnaire and revised for young children. There are 72 items assessing various subscales of parenting behavior.
Change in depression, anxiety, and stress | Change from baseline at 14 weeks and at 3 months
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content.
Satisfaction survey | At treatment completion (approximately 14 weeks after baseline)
  This survey was developed for the Incredible Years and can be found in the Incredible Years manual. It is not standardized.
Weekly IY-ASD evaluation | Weekly throughout treatment (14 weeks total)
  This survey was developed for the Incredible Years and can be found in the Incredible Years manual. It is not standardized.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Dababnah, PhD, Principal Investigator — School of Social Work University of Maryland, Baltimore
Locations (1):
- Onslow County Partnership for Children, Jacksonville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Axberg U, Hansson K, Broberg AG. Evaluation of the Incredible Years Series - an open study of its effects when first introduced in Sweden. Nord J Psychiatry. 2007;61(2):143-51. doi: 10.1080/08039480701226120. PMID 17454729
- [Background] Edwards RT, Ceilleachair A, Bywater T, Hughes DA, Hutchings J. Parenting programme for parents of children at risk of developing conduct disorder: cost effectiveness analysis. BMJ. 2007 Mar 31;334(7595):682. doi: 10.1136/bmj.39126.699421.55. Epub 2007 Mar 9. PMID 17350965
- [Background] Kim E, Cain KC, Webster-Stratton C. The preliminary effect of a parenting program for Korean American mothers: a randomized controlled experimental study. Int J Nurs Stud. 2008 Sep;45(9):1261-73. doi: 10.1016/j.ijnurstu.2007.10.002. Epub 2007 Nov 8. PMID 17996239
- [Background] Webster-Stratton,C. (2011). The Incredible Years: Parents, teachers, and children's training series: Program content, methods, research and dissemination. Seattle, WA: Incredible Years, Inc.
- [Background] Jones K, Daley D, Hutchings J, Bywater T, Eames C. Efficacy of the Incredible Years Basic parent training programme as an early intervention for children with conduct problems and ADHD. Child Care Health Dev. 2007 Nov;33(6):749-56. doi: 10.1111/j.1365-2214.2007.00747.x. PMID 17944785
- [Background] Reid MJ, Webster-Stratton C, Beauchaine TP. Parent training in head start: a comparison of program response among African American, Asian American, Caucasian, and Hispanic mothers. Prev Sci. 2001 Dec;2(4):209-27. doi: 10.1023/a:1013618309070. PMID 11833925
- [Background] Melhuish EC. Parenting training improves problem behaviour in children at risk of conduct disorder. Evid Based Ment Health. 2007 Nov;10(4):125. doi: 10.1136/ebmh.10.4.125. No abstract available. PMID 17962687
- [Background] Smith LE, Seltzer MM, Tager-Flusberg H, Greenberg JS, Carter AS. A comparative analysis of well-being and coping among mothers of toddlers and mothers of adolescents with ASD. J Autism Dev Disord. 2008 May;38(5):876-89. doi: 10.1007/s10803-007-0461-6. PMID 17924181
- [Background] Dababnah S, Parish SL. A Comprehensive Literature Review of Randomized Controlled Trials for Parents of Young Children with Autism Spectrum Disorder. J Evid Inf Soc Work. 2016 May-Jun;13(3):277-92. doi: 10.1080/23761407.2015.1052909. Epub 2015 Jul 15. PMID 26177069
- [Background] Dababnah S, Parish SL. Feasibility of an empirically based program for parents of preschoolers with autism spectrum disorder. Autism. 2016 Jan;20(1):85-95. doi: 10.1177/1362361314568900. Epub 2015 Feb 25. PMID 25717131
- [Background] Dababnah S, Parish SL. Incredible Years program tailored to parents of preschoolers with autism: Pilot results. Research on Social Work Practice 26(4): 372-385. https://doi.org/10.1177/1049731514558004